CLINICAL TRIAL: NCT00034073
Title: Quantitative fMRI in Children and Adults Using Arterial Spin Tagging Techniques
Brief Title: Magnetic Resonance Imaging in Children and Adults Using Arterial Spin Tagging Techniques
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 020182; 02-N-0182
Record Dates: First submitted 2002-04-20; First posted 2002-04-22 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-04-16

CONDITIONS: Healthy
Keywords: Imaging; Pediatrics; Brain; Mapping; Development; Healthy Volunteer; HV; Normal Control

SUMMARY:
This study will use magnetic resonance imaging (MRI) to examine how blood flow to the brain differs at different ages with the brain is at rest, and during performance of tasks that involve language, memory, motor control, and sight. The study will evaluate the usefulness of MRI in identifying language function and location, and may provide information on how the brain develops over time to process brain functions, such as language and memory.

Healthy normal volunteers in three age groups-children 8-10, adolescents 13-16, and young adults 21-30-may be eligible for this study. Participants must be right-handed and be native English speakers. Candidates will be screened via a telephone interview and examination by a neurologist.

Participants will undergo MRI scanning of the brain during rest or while performing a task designed to test a skill. The tasks may involve remembering numbers, reading a word, tapping fingers, or looking at a flashing picture. MRI uses a magnetic field and radio waves to produce pictures of the brain. For the procedure, the subject lies still on a table that is moved into the scanner (a cylinder containing the magnet). Earplugs are worn to muffle loud noises caused by electrical switching of radio frequency circuits used in the scanning process. Adults may spend as long as 90 minutes in the scanner, usually less than 45 minutes. For children, the time is less than 75 minutes-usually 30 to 40 minutes. Participants may be asked to repeat the scans up to 5 times in different sessions to test different brain functions or confirm findings.

DETAILED DESCRIPTION:
FMRI using BOLD technique is an indirect and relative measure of neuronal activity and makes comparison among age groups problematic in light of known age related changes in glucose consumption and resting cerebral blood flow. In this study Arterial Spin Tagging techniques will be used to perform quantitative measures of blood flow changes during fMRI tasks. Children and adults will perform four tasks: primary sensory (photic flash), primary motor (finger tapping), and cognitive (working memory and semantic decision) tasks using parametric block designs, to account for developmental performance, using imaging parameters that allow quantitative measures of cerebral blood flow response as well as BOLD signal. Three age groups will be studied, children 8-10, 14-16, and young adults (21-28). Data will be analyzed using AFNI to identify activated areas. Further analysis will be performed using a region of interest analysis. We will compare quantitative measures at optimal performance levels. The three experimental age groups will be compared for delta rCBF and extent of activated area for each task. The study will determine age dependent changes in blood flow response during cortical activation across ages.

ELIGIBILITY:
* INCLUSION CRITERIA:

Right-handed (Edinburgh Handedness Inventory)

Native English speaker (for language and memory paradigms only)

EXCLUSION CRITERIA:

Medical or technical contraindications to MRI procedures (e.g. no braces, pacemakers, cochlear devices, surgical clips, etc.)

History of neurologic or psychiatric disease or a learning or attentional disorder

One year below grade level

CNS active medications

Pregnancy

Claustrophobia

Inability to comply with the protocol

Volunteers will also be asked if they have a history of dry or irritated eyes and informed this may increase the risk of eye irritation and discomfort in the 3T scanner.

Ages: 8 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70
Dates: Start 2002-04-18; Study Completion 2009-04-16

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Barnes PD. Imaging of the central nervous system in pediatrics and adolescence. Pediatr Clin North Am. 1992 Aug;39(4):743-76. doi: 10.1016/s0031-3955(16)38374-2. PMID 1635805
- [Background] Braver TS, Cohen JD, Nystrom LE, Jonides J, Smith EE, Noll DC. A parametric study of prefrontal cortex involvement in human working memory. Neuroimage. 1997 Jan;5(1):49-62. doi: 10.1006/nimg.1996.0247. PMID 9038284
- [Background] Belliveau JW, Kennedy DN Jr, McKinstry RC, Buchbinder BR, Weisskoff RM, Cohen MS, Vevea JM, Brady TJ, Rosen BR. Functional mapping of the human visual cortex by magnetic resonance imaging. Science. 1991 Nov 1;254(5032):716-9. doi: 10.1126/science.1948051.